CLINICAL TRIAL: NCT05886192
Title: The Construction and Application of Therapeutic System of Intelligent Decision-Oriented Hemodynamic Organized Therapy for Shock Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-PUMCH-B-115
Record Dates: First submitted 2023-05-05; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Septic Shock
Keywords: norepinephrine, vasopressin, organ perfusion.
MeSH Terms: conditions — Shock, Septic; Diabetes Insipidus | interventions — lidocaine, norepinephrine, vasopressin drug combination; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- norepinephrine+vasopressin (Experimental): norepinephrine+vasopressin
  Interventions: Drug: norepinephrine+vasopressin
- Norepinephrine (Placebo Comparator): norepinephrine
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: norepinephrine+vasopressin — Norepinephrine combined with vasopressin to maintain blood pressure
  Arms: norepinephrine+vasopressin
Drug: Norepinephrine — norepinephrine
  Arms: Norepinephrine

SUMMARY:
Patients with septic shock with norepinephrine >0.25ug/kg/min were enrolled. Informed consent was obtained for inclusion in the study and random assignment into the combination or norepinephrine group.

Contact the research assistant to obtain patient number information and print out the appropriate labels.Notify the ward dispensing nurse to open the experimental drug cassette (placed in the refrigerator 4℃ drug cabinet).

Extract the corresponding experimental medication according to the patient label number, dispense it and send it to the ward, label it and hand it over to the bedside nurse to start using it. The time point at which the medication was connected to the patient and activated was recorded as the zero point for the start of the study.

The data were monitored according to the time points specified in the study: baseline,0h , 6h, D1, D2, and post-drug withdrawal.

ELIGIBILITY:
Inclusion Criteria:

Septic shock patients with norepinephrine>0.25ug/kg/min

Exclusion Criteria:

1. Under 18 years of age
2. Acute coronary syndrome requiring treatment
3. have been treated with VA-ECMO
4. VV-ECMO treatment has been administered for less than 12 hours
5. Patient is on posterior pituitary hormone
6. Patients with liver failure with a Model for End-Stage Liver Disease (MELD) score ≥ 30
7. Patients requiring more than 500 mg of hydrocortisone or equivalent glucocorticoid daily as a fixed dose
8. absolute neutrophil counts below 1,000/mm3
9. Patients with active bleeding who are expected to require (within 48 hours of study entry) transfusion of more than 4 units of red blood cell concentrate patients with active bleeding that is expected to require (within 48 hours of study entry) transfusion of more than 4 units of red blood cell concentrate
10. malignancy or other irreversible disease or condition with an estimated 6-month mortality rate of ≥50%
11. Confirmed or suspected acute mesenteric ischemia. If the investigator believes that the patient's condition is highly suspicious but not confirmed by conventional criteria The investigator may exclude a patient if, in the opinion of the investigator, the patient's condition is highly suspicious but not confirmed by conventional criteria, or if the treating physician has initiated empiric therapy.
12. Likely death expected within 12 hours
13. Family or physician plans to implement a palliative care plan for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
28days-Mortality in ICU | 28 days
  28 day mortality rate
ICU duration | an average of 1 year
  Residence time in ICU

SECONDARY OUTCOMES:
RVDEA/LVDEA | baseline,0hour, 6hour, Day1, Day2, and post-drug withdrawal(within 1week)
  bedside cardiac ultrasound parameters,Qualitative indicators: RVDEA/LVDEA
right ventricular thickness | baseline,0hour, 6hour, Day1, Day2, and post-drug withdrawal(within 1week)
  bedside cardiac ultrasound parameters qualitative indicators: right ventricular thickness,
Tricuspid Annular Plane Systolic Excursion | baseline,0hour, 6hour, Day1, Day2, and post-drug withdrawal(within 1week)
  Right ventricular systolic function indicators: Tricuspid,Annular,Plane,Systolic,Excursion (TAPSE) Right ventricular pressure indicators: TV max, peak pulmonary artery regurgitation Other cardiac parameters: E/A, E/E'.
resistance index of superior mesenteric artery | baseline,0hour, 6hour, Day1, Day2, and post-drug withdrawal(within 1week)
  Blood flow parameters of superior mesenteric artery: resistance index 2) VexUS: Liver vein, portal vein, and renal vein. 3) Arterial pressure monitoring waveform. 4) Intestinal ultrasound score
venous excess ultrasound grading system(VexUS) | baseline,0hour, 6hour, Day1, Day2, and post-drug withdrawal(within 1week)
  Liver vein, portal vein, and renal vein.
Intestinal ultrasound score | baseline,0hour, 6hour, Day1, Day2, and post-drug withdrawal(within 1week)
  Intestinal ultrasound score :Including the diameter of the small intestine, the thickness of the small intestine wall, and the frequency of small intestine peristalsis
pulsatility index of the middle cerebral artery | baseline,0hour, 6hour, Day1, Day2, and post-drug withdrawal(within 1week)
  Cranial ultrasound measurement indexes Cranial ultrasound measurement indexes: pulsatility index of the middle cerebral artery

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No